CLINICAL TRIAL: NCT04968496
Title: Isolating Food Insecurity to Understand Childhood Health Outcomes and Biological Mechanisms of Risk
Brief Title: Biobehavioral Mechanisms of Food Insecurity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study PI has resigned
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1773080
Record Dates: First submitted 2021-06-15; First posted 2021-07-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-10

CONDITIONS: Food Insecurity; Obesity, Childhood; Inflammation; Mental Health
MeSH Terms: conditions — Pediatric Obesity; Inflammation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Insecure Group (No Intervention): Children randomized to the naturally-occurring Food Insecure group will receive a weekly newsletter with information on available area-specific food programs. The weekly newsletter will be sent in two ways: 1) a paper copy will be mailed and 2) a link to an electronic version will be sent via Ilumivu to families to remove any barriers to engagement with the information. In the absence of school meal programs, children from low-income households are at increased risk for food insecurity during the summer.37-39 Given low engagement in summer food programs, it is not expected that this newsletter will impact food security in this group.
- Food Secure Group (Experimental): Children randomized to the Food Secure group will receive breakfast and lunch meals for eight weeks throughout the summer. Weekly meals will be delivered to each participant's home by Yumble, a company that prepares meals for children ages 3 to 12 years and ships them fresh in insulated, food safe packaging to the home. The meals have similar nutrition standards to those offered via the National School Lunch Program and include fruits, vegetables, whole grains, and lean/ vegetarian proteins. To accommodate cultural preferences or dietary constraints, Yumble offers 20 different breakfast, lunch and dinner meals each week. Families will choose their weekly menus to improve adherence. Participants who have siblings in their home will be provided a family meal kit, which provides 24 meals each week. Additional meals will help to prevent household food insecurity and ensure that the child enrolled in the study consumes the meals each week.
  Interventions: Other: Food Secure Group

INTERVENTIONS:
Other: Food Secure Group — Weekly meals (five breakfast and five lunch meals) will be provided to all children randomized to this group to prevent the onset of summertime food insecurity
  Arms: Food Secure Group

SUMMARY:
Food insecurity is prevalent in the United States. Defined as unstable and inadequate access to food, food insecurity disproportionately affects low-income households, those with children and those with a Black or Hispanic head of household. Moreover, food insecurity is associated with childhood obesity, a relationship that is not well understood from a behavioral or biological perspective. This randomized controlled trial will take advantage of the natural onset of summertime food insecurity among school-age children, ages 8-12 years, to examine the biobehavioral mechanisms of food insecurity including diet quality, biomarkers of Metabolic Syndrome, inflammation, and stress, weight status, and measures of child mental health.

DETAILED DESCRIPTION:
Food insecurity affects one in six households with children in the United States and disproportionately impacts those headed by women and minorities. Food insecurity is associated with childhood obesity, asthma, anxiety and depression and behavioral problems, and thus contributes to health disparities. While food insecurity likely contributes to poor health through its effect on diet, such a simplistic understanding likely obscures the effects of stress - those unique to childhood, such as Adverse Childhood Experiences including maternal depression, as well as those generally associated with the experience of poverty. To inform the mechanisms by which food insecurity ultimately affects physical and mental health outcomes in children, this study will disentangle the effects of food insecurity from those of poverty and examine effects on diet, biomarkers, weight gain, mood and behavior while considering other childhood adversities. Specifically, through a unique summertime meal provision intervention, the proposed project will isolate the experience of food insecurity in children, ages 8 to12 years, from low-income households in Providence, RI. In partnership with the YMCA of Greater Providence and the Healthy Communities Office in Providence, we will recruit 100 children over two summers. After completing a baseline assessment, participants will be randomized to receive home-delivered meals throughout the summer or to receive a weekly newsletter. Children randomized to the newsletter group will experience the natural onset of summertime food insecurity and receive a weekly newsletter on community resources that is not expected to affect food insecurity (Food Insecure Group). Those randomized to receive meals will remain food secure over the summer through receipt of weekly shipments of five breakfast and lunch meals that meet the nutrition needs of this age group (Food Secure Group). Primary endpoints include diet quality, biomarkers of Metabolic Syndrome, inflammation, and stress, BMI z-scores, and child measures of behavior and anxiety and depression symptoms. The impact of caregiver mood and stress on the health effects of food insecurity will also be explored. Ultimately, findings from this research will clarify the mechanisms by which food insecurity affects child health outcomes and inform how to more effectively prevent food insecurity.

ELIGIBILITY:
Inclusion Criteria:

* ability of parent and child to speak, read and write English or Spanish
* agreement to study participation and random assignment.

Exclusion Criteria:

* Children will not be eligible if they are enrolled in a full-time camp, day care or programming in which regular meals are provided for more than one-week over the summer.
* Children will not be eligible if their Parent / caregiver does not have reliable phone access to complete study measures.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Dietary Quality | 2 months
  Healthy Eating Index (HEI 2015) - scores range from 0 to 100, with 100 representing perfect adherence to the Dietary Guidelines for Americans, 2015
Markers of Inflammation | 3 months
  Blood sample analyzed for C-reactive protein
Markers of Inflammation | 3 months
  Blood sample analyzed for interleukin-6 levels
Markers of Metabolic Syndrome | 3 months
  Blood sample analyzed for glucose
Markers of Metabolic Syndrome | 3 months
  Blood sample analyzed for hemoglobin A1c
Markers of Metabolic Syndrome | 3 months
  Blood sample analyzed for insulin
Markers of Stress | 3 months
  Blood sample analyzed for cortisol
Markers of Stress | 3 months
  Blood sample analyzed for leptin
Markers of Stress | 3 months
  Blood sample analyzed for adiponectin
Child Mood | 3 months
  PROMIS (Patient-Reported Outcomes Measurement Information System) short-form measures for assessing anxiety in children. Scores range from 10 to 50 with a higher score indicating greater anxiety symptoms.
Child Mood | 3 months
  PROMIS (Patient-Reported Outcomes Measurement Information System) short-form measures for assessing depression in children. Scores range from 0 to 32 with a higher score indicating greater depressive symptoms.
Child weight status | 3 months
  Body Mass Index z-score (BMIz) - Z-score will be determined based on child's BMIz for age and sex using the CDC growth charts

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Housing Authority, Newport, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans EW, Jelalian E, Dunsiger S, Villalta D, Tyrka A. Design of a clinical trial to isolate the experience of food insecurity and elucidate the biological mechanisms of risk for childhood health outcomes. Contemp Clin Trials. 2022 Jun;117:106751. doi: 10.1016/j.cct.2022.106751. Epub 2022 Apr 2. PMID 35381377